CLINICAL TRIAL: NCT06891612
Title: Etude Par électroencéphalographie Des mécanismes d'Inhibition de Souvenirs émotionnels Chez le Sujet Jeune Sain
Brief Title: Electroencephalographic Study of the Mechanisms of Inhibition of Emotional Memories in Young Healthy Subjects
Acronym: ENGRAMME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C15-70
Record Dates: First submitted 2025-03-12; First posted 2025-03-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-03

CONDITIONS: Anxiety; Depression; Cognitive Control
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Eye-Tracking Technology; Electroencephalography; Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- pretest healthy participants (Experimental)
  Interventions: Behavioral: Cognitive Assessments; Device: Eye-tracking; Device: Electroencephalography (EEG); Device: Electrocardiography (ECG)
- healthy participant 10 min delayed recall (Experimental): 10 min delayed recall
  Interventions: Behavioral: Cognitive Assessments; Device: Eye-tracking; Device: Electroencephalography (EEG); Device: Electrocardiography (ECG)
- healthy participant 24 h delayed recall (Experimental): 24 h delayed recall
  Interventions: Behavioral: Cognitive Assessments; Device: Eye-tracking; Device: Electroencephalography (EEG); Device: Electrocardiography (ECG)

INTERVENTIONS:
Behavioral: Cognitive Assessments — Cognitive Assessments
Device: Eye-tracking — measurement of the points of gaze
Device: Electroencephalography (EEG) — Electrophysiological monitoring method to record electrical activity of the brain
Device: Electrocardiography (ECG) — measurement of the electrical activity of the heart

SUMMARY:
Forgetfulness has long been considered a pathology of memory. However, the brain's voluntary suppression of certain unpleasant memories is essential for building a healthy memory. This suppression capacity can be measured using the "Think/No-Think" (TNT) paradigm.However, while the areas involved in these processes of suppression are now well described, the nature and temporal dynamics of the processes of inhibition and orientation of attention is still poorly defined. The aim of this study is to describe the nature of the attentional and inhibitory mechanisms involved in the suppression of emotionally negative memories, and their temporal articulation using electroencephalography (EEG). To this end, we will use a model of memory deletion derived from a perceptual attentional task and simulating the deletion phase in order to control the nature and timing of the processes involved. This approach will allow us to observe the presence of correspondences between the responses measured during the attentional test simulating the suppression and the actual phase of suppression, for which we cannot control the nature of the operations undertaken by the subject. In addition, we will assess the emotional response through physiological measures of autonomic nervous system activity (heart rate and electrodermal response) immediately after the TNT phase or one day later, which will allow us to evaluate the influence of memory suppression mechanisms on their emotional content.

From a practical point of view, this study is organized into 3 groups of participants (healthy young adults). Each group will perform a perceptual attentional test and a TNT task, which will be preceded and followed by a measure of emotional response. Group 1 will allow us to test our main hypothesis from a behavioral point of view, as well as to calibrate the attentional task and its consistency with the TNT task. Group 2 will carry out the same tests but during an EEG examination to decode the temporal dynamics of attention states during the process of memory suppression. Group 3 will perform these same tests with a 24-hour interval between the TNT phase and the emotional assessment to estimate the effect of a retention period on forgetfulness functions.

The description of these mechanisms and their physiological correlates will allow us to better understand how this ability to voluntarily control the flow of thoughts associated with negative memories is implemented, and thus to better understand the alterations in this capacity that can be observed during certain mental pathologies such as anxiety or depression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 35 years
* Affiliated to a social security scheme
* Having French as their mother tongue
* Right-handed
* High school graduate or equivalent
* Having signed a written informed consent

Exclusion Criteria:

* Pregnancy in progress, pregnancy test will be performed
* Person deprived of liberty by judicial or administrative decision
* Person hospitalized without consent and not subject to legal protection measures, and person admitted to a health or social care facility for purposes other than research
* Minor
* Adults subject to legal protection measure (guardianship, curatorship or judicial protection), adults unable to express their consent and not subject to protection measure
* Person subject to an exclusion for another research
* History of a neurological, psychiatric disorders, or head trauma with loss of consciousness for more than an hour
* History of cancer over the last 5 years, with the exception of squamous cell carcinomas of the skin
* Presence or history of chronic alcoholism or drug addiction
* Taking medications that may alter cognitive and/or brain function (decision of the principal investigator)
* Presence of visual and/or auditory disorders sufficiently significant to affect the progress of the tests
* Contraindications to electroencephalography
* Presentation of unpleasant images that are too emotionally disturbing for the participant (by decision of the physician)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Completion psychopathological scales | Inclusion visit
  Entered into a computer
Measurement of the electrodermal conductance | Day1
  For emotional evaluation when presenting negative images
Measuremet of heart rate | Day 1
  For emotional evaluation when presenting negative images

SECONDARY OUTCOMES:
Attentional task | Day 1 and Day 2
  This test is performed on a computer after learning pairs of images
Test of "Think/No-Think" | Day1 and Day2
  This test is performed on a computer after learning pairs of images
Measurement of the electrodermal conductance | Day 1 and Day 2
  For emotional evaluation after learning pairs of images
Measuremet of heart rate | Day 1 and Day 2
  For emotional evaluation after learning pairs of images
Measurement of electroencephalographic activity | Day1 and Day 2
  Subjects will be equiped with electrodes during the attentional task and " Think/No-Think " test

CONTACTS AND LOCATIONS:
Locations (1):
- Service de neurologie CHU de Caen, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Legrand N, Etard O, Vandevelde A, Pierre M, Viader F, Clochon P, Doidy F, Peschanski D, Eustache F, Gagnepain P. Long-term modulation of cardiac activity induced by inhibitory control over emotional memories. Sci Rep. 2020 Sep 14;10(1):15008. doi: 10.1038/s41598-020-71858-2. PMID 32929105